CLINICAL TRIAL: NCT07242937
Title: Cultural Intelligence and Learning in Virtual Reality: How Cultural Background Shapes Cognitive and Motor Adaptation
Brief Title: How Cultural Background Affects Cognitive and Motor Learning Using Virtual Reality
Status: Completed | Type: Observational
Sponsor: Bahçeşehir University (Other)
Collaborators: CogniFit Limited (Unknown)
Responsible Party: Principal Investigator, Yara Atef Skout, Principal investigator, Bahçeşehir University
Other Study IDs: E-10840098-202.3.02-5347
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Function; Neuroplasticity; Motor Skills; Virtual Reality; Cross-Cultural Comparison

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Home Group: Participants who lived for at least ten years in their home country with no long-term intercultural exposure. All participants followed the same standardized assessment procedure, including cognitive testing, motor coordination testing, and virtual reality (VR) task performance. No interventions were assigned; the study compared natural learning differences between pre-existing cultural groups.
  Interventions: Behavioral: Virtual reality beat saber training and cognitive and motor assessment
- Abroad group: Participants who lived abroad for at least ten years with long-term intercultural exposure. All participants completed the same standardized assessment procedure, identical to the Home group. No experimental intervention or assignment occurred.
  Interventions: Behavioral: Virtual reality beat saber training and cognitive and motor assessment

INTERVENTIONS:
Behavioral: Virtual reality beat saber training and cognitive and motor assessment — All participants completed the same four-day assessment procedure consisting of cognitive evaluation (Cognitive Assessment Battery-Professional [CAB PRO]), fine-motor coordination testing (Purdue Pegboard Test), and performance on a virtual reality (VR) Beat Saber task using the Meta Quest 2 headset. These procedures were administered equally to all participants. No interventions were assigned; the study observed natural performance differences between pre-existing cultural groups.

SUMMARY:
This observational study examined how long-term cultural background is associated with differences in cognitive and motor learning within a virtual reality environment. Forty-three healthy university students participated in four days of standardized assessment procedures involving cognitive testing, fine-motor evaluation, and performance on a virtual reality (VR) task. Participants were classified into two pre-existing groups based on long-term cultural exposure: a Home group (lived mainly in their native country) and an Abroad group (lived abroad for at least ten years). All participants completed the same assessment procedures. The study observed natural variations in cognitive performance, motor coordination, and VR learning progression across sessions.

DETAILED DESCRIPTION:
This observational study examined how long-term cultural background is associated with differences in cognitive and motor learning within a virtual reality (VR) environment. The study used a case-control design based on naturally existing groups. Participants were not assigned to conditions. Instead, they were classified into two groups according to their long-term cultural exposure: a Home group (lived primarily in their native country for at least ten years) and an Abroad group (lived abroad for at least ten years).

All participants followed the exact same schedule and attended the study sessions on four fixed days: Monday, Wednesday, Friday, and the following Monday. This controlled scheduling ensured that all participants experienced the same time intervals between sessions, eliminating variability due to inconsistent spacing.

During Day 1, participants completed baseline assessments, including:

CogniFit cognitive battery, evaluating attention, memory, processing speed, and executive functions

Purdue Pegboard Test, assessing fine-motor coordination

IFIS scale (Index of Fit Self-Perception) to assess physical fitness

Cultural Intelligence Scale (CQS) to measure cultural intelligence

After completing the baseline assessments on Day 1, participants performed the standardized VR learning task (Beat Saber).

On Days 2 and 3 (Wednesday and Friday), participants completed only the VR Beat Saber task. These sessions were used to measure progression of visuomotor learning, accuracy, speed, and performance over time.

On Day 4 (the following Monday), participants again completed:

CogniFit cognitive battery

Purdue Pegboard Test

The VR Beat Saber task

Repeating these tests on Day 4 allowed the study to evaluate changes in cognitive performance and motor coordination across the study period, as well as overall VR learning progression.

All procedures and assessments were identical for both groups. The study did not manipulate behavior or deliver interventions; instead, it observed naturally occurring differences in learning and performance across participants with different long-term cultural backgrounds. This design allowed the analysis of how cultural exposure may relate to cognitive adaptation, motor learning, and VR-based task progression. No biospecimens were collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy university students aged 17-35
* Lived at least ten years in either their home country (Home group) or abroad (Abroad group)
* Fluent in English
* Normal or corrected-to-normal vision
* Able to use virtual reality headset and controllers
* Provided informed consent

Exclusion Criteria:

* History of neurological or psychiatric disorders
* Severe visual or motor impairment
* Use of medications affecting cognition
* Any condition preventing safe participation in VR tasks

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy university students aged 17-35. Participants were divided into two cohorts based on long-term cultural exposure: Home group (lived in their home country for at least ten years) and Abroad group (lived abroad for at least ten years). All participants were fluent in English and completed four days of cognitive assessments and VR gameplay sessions.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Cognitive Performance Score (CogniFit CAB PRO) | Day 1 and Day 4
  Computerized cognitive assessment measuring attention, memory, reasoning, and executive functions. Composite cognitive score is calculated using the Cognitive Assessment Battery-Professional [CAB PRO]) battery.

SECONDARY OUTCOMES:
Motor Dexterity (Purdue Pegboard Test) | Day 1 and Day 4
  Fine-motor coordination assessed using the Purdue Pegboard Test, including dominant hand, non-dominant hand, both hands, and assembly scores.
VR Gameplay Accuracy (Beat Saber Cut Accuracy) | Day 1 to Day 4
  Percentage of targets cut correctly during Beat Saber gameplay, reflecting visuomotor precision and learning progression.
VR Gameplay Performance (Beat Saber Combo Length) | Day 1 to Day 4
  Maximum consecutive successfully hit targets ("combo streak") recorded during each virtual reality session to evaluate learning and consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Gözener Canbülbül, Study Director — Bahçeşehir University
Locations (1):
- Bahcesehir University- Faculty of Health Sciences, Istanbul, Turkey (Türkiye)